CLINICAL TRIAL: NCT05971940
Title: A Phase 3, Randomized, Double-Blind Study to Investigate the Efficacy and Safety of Once Daily Oral LY3502970 Compared With Placebo in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise Alone
Brief Title: A Study of Orforglipron (LY3502970) in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise Alone
Acronym: ACHIEVE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18564; J2A-MC-GZGT (Other: Eli Lilly and Company); U1111-1290-5157 (Other: UTN Number)
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally.
  Other Names: LY3502970
  Arms: Orforglipron Dose 1; Orforglipron Dose 2; Orforglipron Dose 3
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine safety and efficacy of orforglipron compared with placebo in adult participants with type 2 diabetes and inadequate glycemic control with diet and exercise alone. The study will last approximately 54 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes
* Have HbA1c ≥7.0% (53 mmol/mol) to ≤9.5% (80 mmol/mol) despite diet and exercise treatment, as determined by the central laboratory at screening.
* Are naïve to insulin therapy except for gestational diabetes or ≤14 days use for acute treatment and have not used any oral or injectable antihyperglycemic medications during the 90 days preceding screening or between screening and randomization.
* Are of stable weight (±5%) for at least 90 days prior to screening and agree to not initiate an intensive diet or exercise program during the study with the intent of reducing body weight other than the lifestyle and/or dietary measures for diabetes treatment.
* Have a body mass index (BMI) ≥23.0 kilogram/square meter (kg/m²) at screening.

Exclusion Criteria:

* Have Type 1 Diabetes
* Have a history of ketoacidosis or hyperosmolar state or coma within the last 6 months prior to screening, or between screening and randomization.
* Currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema
* Have New York Heart Association functional classification IV congestive heart failure.
* Have acute or chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 40

SECONDARY OUTCOMES:
Percentage of Participants with an HbA1c target value of <7.0% (53 mmol/mol) | Week 40
Percentage of Participants with an HbA1c target value of ≤6.5% (48 mmol/mol) | Week 40
Change from Baseline in Fasting Serum Glucose | Baseline, Week 40
Percentage Change from Baseline in Body Weight | Baseline, Week 40
Change from Baseline in Body Weight | Baseline, Week 40
Change from Baseline in Daily Average 7-point Self-Monitored Blood Glucose (SMBG) | Baseline, Week 40
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 40
Change from Baseline in Non-HDL Cholesterol | Baseline, Week 40
Percentage Change from Baseline in Triglycerides | Baseline, Week 40
Percentage of Participants Who Achieved Weight Loss of ≥5% | Week 40
Change from Baseline in Short Form 36 Version 2 (SF-36v2) Acute Form Domain Scores | Baseline, Week 40

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (89):
- United States (41):
  - Syed Research Consultants Llc, Sheffield, Alabama
  - Epic Medical Research - Surprise, Surprise, Arizona
  - Quality of Life Medical & Research Center, Tucson, Arizona
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Ark Clinical Research, Long Beach, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Infinity Clinical Research - Norco, Norco, California
  - Norcal Endocrinology & Internal Medicine, San Ramon, California
  - University Clinical Investigators, Inc., Tustin, California
  - Connecticut Clinical Research - Cromwell, Cromwell, Connecticut
  - Invictus Clinical Research Group, Coconut Creek, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - K2 Medical Research, Maitland, Florida
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Family First Medical Center, Idaho Falls, Idaho
  - American Health Network of Indiana, LLC - Muncie, Muncie, Indiana
  - Tekton Research - Wichita, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Revival Research Institute, Dearborn, Michigan
  - Billings Clinic, Billings, Montana
  - Ellipsis Research Group - Brooklyn - 7th Street, Brooklyn, New York
  - Central New York Clinical Research, Manlius, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lucas Research - New Bern, New Bern, North Carolina
  - Centricity Research Dublin Multispecialty, Dublin, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - The Research Center of The Upstate, Greenville, South Carolina
  - MDFirst Research, LLC, Lancaster, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Juno Research, Houston, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - Amir A Hassan, MD, PA, Houston, Texas
  - Burke Internal Medicine and Research, Burke, Virginia
- China (15):
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Luhe Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Pinggu District Hospital, Beijing, Beijing Municipality
  - Shunde Hospital of Southern Medical Univesity, Foshan, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Nanyang First People's Hospital, Nanyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Jinan, Shandong
  - Pudong New Area People's Hospital Shanghai, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
- India (9):
  - GMERS Medical College and General Hospital, Vadodara, Gujarat
  - M S Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Medstar Speciality Hospital, Bangalore, Karnataka
  - BSES MG Hospital, Mumbai, Maharashtra
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur, Maharashtra
  - Grant Medical Foundation - Ruby Hall Clinic, Pune, Maharashtra
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Kumudini Devi Diabetes Research Center, Hyderabad, Telangana
  - Institute of Post Graduate Medical Education and Research and Seth Sukhlal Karnani Memorial Hospital, Kolkata, West Bengal
- Japan (14):
  - Tokuyama Clinic, Mihama-ku,Chiba City, Chiba
  - Steel Memorial Yahata Hospital, Kitakyushu, Fukuoka
  - Hasegawa Medical Clinic, Chitose, Hokkaido
  - MinamiAkatsukaClinic, Mito, Ibaraki
  - Iwamoto Clinic, Zentsujichó, Kagawa-ken
  - Hayashi Diabetes Internal Medicine Clinic, Chigasaki, Kanagawa
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - The Institute of Medical Science, Asahi Life Foundation, Chuo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku, Tokyo
  - Morinaga Ueno Clinic, Kumamoto
  - Abe Clinic, Ōita
- Mexico (8):
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occidente, Guadalajara, Jalisco
  - Centro de Investigacion Medica Integral, Guadalajara, Jalisco
  - Salud Cardiovascular, Guadalajara, Jalisco
  - Centro de Investigacion Medica de Occidente, S.C., Zapopan, Jalisco
  - Investigacion En Salud Y Metabolismo S.C / Nutricion Clinica / Unidad de Base de Datos, Chihuahua City
  - PanAmerican Clinical Research - Querétaro - Avenida Antea, Querétaro
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
  - FAICIC S. de R.L. de C.V., Veracruz
- Puerto Rico (2):
  - Puerto Rico Health Institute, Dorado
  - Advance Medical Research Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Rosenstock J, Hsia S, Nevarez Ruiz L, Eyde S, Cox D, Wu WS, Liu R, Li J, Fernandez Lando L, Denning M, Ludwig L, Chen Y; ACHIEVE-1 Trial Investigators. Orforglipron, an Oral Small-Molecule GLP-1 Receptor Agonist, in Early Type 2 Diabetes. N Engl J Med. 2025 Sep 18;393(11):1065-1076. doi: 10.1056/NEJMoa2505669. Epub 2025 Jun 21. PMID 40544435
- See also: A Study of Orforglipron (LY3502970) in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise Alone (ACHIEVE-1) — https://trials.lilly.com/en-US/trial/413375